CLINICAL TRIAL: NCT06442852
Title: Study on the Relationship Between Peripheral Blood miRNA and Risk and Severity of Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Jiajie Chen (Other)
Responsible Party: Sponsor-Investigator, Jiajie Chen, doctor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20210116
Record Dates: First submitted 2024-05-30; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; MicroRNAs
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimer's disease patients: Alzheimer's patients who meet the inclusion criteria and sign an informed consent form
  Interventions: Other: exposure
- Healthy control: Healthy volunteers who meet the inclusion criteria and sign informed consent
  Interventions: Other: exposure

INTERVENTIONS:
Other: exposure — The observed exposure factor was the expression level of synaptic associated mirna in the serum of patients with Alzheimer's disease and healthy volunteers

SUMMARY:
Alzheimer's Disease, AD is a type of neurofibrillary tangles formed by the deposition of beta amyloid proteins within the nervous system cells and excessive phosphorylation of extracellular Tau proteins, NFTs are the main pathological features of central nervous system degeneration, also known as senile dementia. In addition, synaptic plasticity damage and neuroinflammation also play important roles in the progression of AD. Neurosynapses are the sites where neurons interact with each other in terms of function, and are also crucial for neuronal information transmission and communication. Synapses are the fundamental units in the brain, and synaptic activity can stimulate the maturation of mushroom like dendritic spines and form new synapses, enabling synaptic strength to adapt to changes in the internal and external environment, thereby playing an important role in learning and memory. Previous studies have shown that synaptic activity interruption and synaptic loss can already be detected in the AD brain, especially in the early stages. Multiple studies have shown a higher correlation between synaptic disorders characterized by synaptic loss and decreased synaptic activity and cognitive impairment in Alzheimer's disease compared to age-related plaques and neurofibrillary tangles. Therefore, understanding the potential mechanisms of synaptic disorders will contribute to the development of early treatment strategies for AD. MicroRNAs (miRNAs) are a type of small non coding RNA with a length of approximately 22 nucleotides. Their main function is to silence target genes at the post transcriptional level and inhibit the translation process of their proteins. MiRNAs are involved in many physiological processes and pathological pathways, including development, tumorigenesis, and heart disease. Recently, people have also studied the abnormal regulatory role of miRNAs in AD synaptic disorders. Some miRNAs enriched in the brain, such as miR-124, MiR-132 is abnormally expressed in the AD brain, mediating synaptic plasticity damage. However, most of the miRNAs mentioned above are not directly related to synaptic activity, and their regulation of AD synaptic damage is likely to be a broad-spectrum effect. At present, there are 12 miRNAs closely related to synaptic plasticity that have been identified. By detecting changes in miRNAs closely related to synaptic plasticity in peripheral blood of AD patients and healthy volunteers, and exploring their relationship with the severity of AD lesions, it may provide new directions for early diagnosis of AD. The purpose of this study is to: (1) detect the expression levels of miRNAs closely related to synaptic plasticity in the peripheral blood of healthy volunteers and AD patients, and identify the miRNAs with the greatest differences; (2) Analyze the relationship between the expression levels of the aforementioned miRNAs in the peripheral blood of AD patients and the severity of the disease; (3) Analyze the relationship between the expression levels of the aforementioned miRNAs in the peripheral blood of AD patients and the commonly used neuropsychiatric scale scores. We plan to clarify the changes in peripheral blood miRNAs and their relationship with the severity of AD through case-control studies, in order to provide new directions for early diagnosis of AD.

ELIGIBILITY:
Inclusion Criteria:

Alzheimer's disease patients:

* Meet the diagnostic criteria of NINCDS-ADRDA for AD
* Clinical Dementia Scale (CDR) score ≥0.5

Healthy volunteers:

* No complaints or symptoms of cognitive impairment
* MMSE score is higher than the threshold value

Exclusion Criteria:

Alzheimer's disease patients:

* Dementia or cognitive impairment due to other diseases
* Combined with delirium
* A history of drug abuse
* Severe deafness, aphasia and other impact scale score

Healthy volunteers:

* had an organic brain lesion
* Suffering from other major physical diseases: such as severe immune diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Alzheimer's patients or healthy volunteers at Tongji Hospital in Wuhan
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
miR-135a | December 2024
  synaptic associated miRNA

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zheng, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China